CLINICAL TRIAL: NCT04370262
Title: A Multi-site, Randomized, Double-Blind, Comparative Trial of the Safety and Efficacy of Standard of Care (SOC) Plus Famotidine vs SOC Plus Placebo for the Treatment of COVID-19 in Hospitalized Adults
Brief Title: Multi-site Adaptive Trials for COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Joseph Conigliaro, Vice Chairperson, Medicine, General Internal Medicine, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-0268
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
Keywords: COVID-19; Coronavirus; Famotidine
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind Comparative Trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SOC/Famotidine (Active Comparator): Subjects in this study arm will receive a combination of Standard of Care (SOC) treatment and intravenous famotidine. Famotidine Injection, 10mg/mL mixed with Normal Saline is given intravenously at 120mg (30% of 400 mg oral dose). The total daily dose proposed is 360mg/day famotidine IV for a maximum of 14 days, or hospital discharge, whichever comes first. SOC will be administered as per the current clinical protocol for COVID-19.
  Interventions: Drug: SOC + Intravenous Famotidine
- SOC/Placebo (Placebo Comparator): Subjects in this arm will receive the current Standard of Care treatment for COVID-19; plus placebo infusion three times daily.
  Interventions: Drug: SOC + Placebo

INTERVENTIONS:
Drug: SOC + Intravenous Famotidine — Standard of Care treatment plus IV famotidine
  Arms: SOC/Famotidine
Drug: SOC + Placebo — Standard of Care treatment plus IV placebo
  Arms: SOC/Placebo

SUMMARY:
The overall objective of the study is to evaluate the clinical efficacy of COVID-19 treatments consisting of standard of care (SOC), vs SOC with high dose famotidine in patients hospitalized and meeting radiologic criteria for COVID-19 disease. SOC for the treatment for COVID-19 has evolved since the initial conceptualization of this protocol and early recruitment of patients. Initially SOC included hydroxychloroquine and has progressed to include Remdesivir. This protocol is amended to allow the SOC to reflect the prevailing treatment for COVID-19. We will compare clinical outcomes associated with SOC and the addition of high-dose intravascular famotidine. The trial is designed to enroll at least 471 COVID-19 patients hospitalized with moderate to severe disease into each of the two treatment arms, with a total enrollment target of at least 942 patients. This trial has been designed and powered to support up to three interim analyses that will enable prompt assessment of benefits and risks of the two treatment groups while maintaining the rigorous gold standard of a randomized double blind clinical trial structure. Trial design has been guided by practical consideration of the current clinical context involving rapidly escalating demands on hospital staff and resources, and incorporates a minimalist approach employing existing laboratory information management systems and a clinically relevant binary primary outcome of 30-day endpoint of death or survival.

DETAILED DESCRIPTION:
In December 2019, the Wuhan Municipal Health Committee identified an outbreak of viral pneumonia cases of unknown cause. Coronavirus RNA was quickly identified in these patients. This novel coronavirus has been designated SARS-CoV-2, and the disease caused by this virus has been designated COVID-19 and has infected hundreds of thousands of confirmed individuals in more than 200 countries. Currently there are no approved therapeutic agents available for coronaviruses. There is an urgent need for an effective treatment to treat symptomatic patients but also to decrease the duration of virus transmission in the community. Among candidate drugs to treat COVID-19, repurposing of FDA-approved drugs for use as antiviral treatments is proposed because knowledge on safety profile, side effects, and drug interactions are well known.

In silico screening of FDA licensed compound libraries against the SARS CoV 2 protease Plpro catalytic site was performed using solved crystal structures of the protein. Plpro (Papain-like protease) is an early acting protease responsible for initial processing of the SARS CoV2 polyprotein into active subunits. Plpro also has ubiquitinase activity, and is implicated in early infection phase inhibition of innate (interferon) immune responses which otherwise would suppress viral replication. A ranked list of licensed compounds with predicted binding activity in the Plpro catalytic site was computationally generated, and the Plpro catalytic site binding pose of each of the top compounds was examined and ranked by a team of pharmaceutical chemists. Package inserts or product monographs for the licensed compounds which generated high computational binding scores and passed inspection were then reviewed and used to rank compounds based on adverse events, warnings, drug interactions on-target mechanisms, pharmacokinetic and absorption, metabolism, excretion and toxicity (ADMET), protein binding and available therapeutic window considerations. Famotidine (Pepcid), a histamine H2 antagonist widely available over-the-counter, was repeatedly computationally scored among the highest of the compounds tested, and was associated with the most favorable pharmacokinetic and safety profile. A series of analogs of famotidine were generated using PubChem, and many of these scored even higher as potential candidates. This control compound set further confirmed the predicted binding of the molecular backbone chemotype at the Plpro protease/ubiquitinase site. Currently available as oral and IV products, famotidine has a very attractive proven safety, drug interaction, and therapeutic window profile. Samples of famotidine have been submitted at Southern Research and IITRI for in vitro testing in COVID-19 cultures. Unpublished anecdotal case studies suggest clinical benefits associated with administration of famotidine 40 mg PO TID in mild COVID-19 infection.

On 29 April 2020, the National Institute of Allergy and Infectious Diseases (NIAID) announced that Remdesivir was better than placebo in reducing time to recovery for people hospitalized with advanced COVID-19 and lung involvement. In an earlier study of adult patients admitted to a hospital for severe COVID-19, Remdesivir was not associated with statistically significant clinical benefits. In that study, Remdesivir was not associated with a difference in time to clinical improvement. Although not statistically significant, patients receiving Remdesivir had a numerically faster time to clinical improvement than those receiving placebo among patients with symptom duration of 10 days or less. Remdesivir was stopped early because of higher numbers of adverse events compared to placebo. Because of these studies the FDA stated on 1 May 2020, that it is "reasonable to believe" that known and potential benefits of Remdesivir outweigh its known and potential risks, in some specific populations hospitalized with severe COVID-19.

Given the refinement of standard of care to include Remdesivir and no longer hydroxychloroquine, we have edited the study protocol to reflect this new standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
2. Understands and agrees to comply with planned study procedures.
3. Male or non-pregnant female adult ≥18 years of age at time of enrollment.
4. Subject consents to randomization within 36 hours of hospital admission.
5. Has radiographic confirmed COVID-19 disease < 72 hours prior to randomization.
6. Illness of any duration, and at least one of the following:

   * Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), OR
   * Clinical assessment (evidence of rales/crackles on exam) AND SpO2 ≤ 94% on room air, OR
   * Requiring mechanical ventilation and/or supplemental oxygen.
7. Subjects do not require laboratory confirmation of the corona virus SARS-CoV-2 to determine eligibility
8. Women of childbearing potential must agree to use at least one primary form of contraception for the duration of the study (acceptable methods will be determined by the site).

Exclusion Criteria:

1. Mild COVID-19 disease (minor clinical symptoms, imaging does not show signs of lung inflammation)
2. Recent history of or any in-hospital exposure to investigational medications targeting COVID-19, or concurrent participation in a clinical trial targeting COVID-19
3. ALT/AST > 5 times the upper limit of normal.
4. Moderate renal insufficiency (creatinine clearance 30-50 mL/min) OR Stage 4 severe chronic kidney disease OR requiring dialysis (i.e. creatinine clearance <30 mL/min)
5. History of or evidence of QT prolongation on ECG examination
6. History of psoriasis or porphyria
7. Absolute neutrophil count (ANC) is < 2000 mm3
8. Pregnancy
9. History of hepatic disease, Hepatitis C infection, or alcoholism
10. History of G-6-PD (glucose-6-phosphate dehydrogenase) deficiency
11. Concomitant use of the following medications: atazanavir, dasatinib, neratinib, ozanimod, pazopanib, rilpivirine, siponimod, and/or tizanidine.
12. Anticipated transfer to another hospital which is not a study site within 72 hours.
13. Allergy to any study medication
14. Known to be immunocompromised by disease or treatment for existing disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days post hospitalization
  Mortality status

SECONDARY OUTCOMES:
Virologic response to study treatment detected in blood | Day 30 relative to admission Day 0
  Percent change in PCR copy number from first measurement
Virologic clearance in nasal swab and/or lower respiratory secretions | Day 6 and Day 30
  Presence or absence of SARS-CoV-2 Viral RNA in Nasopharyngeal swab or lower respiratory secretions
Clinical Severity | Measured on study Days 3, 5, 8, 11, 15 and 30.
  Measured by 7-point ordinal scale: from (1) death, to (7) not hospitalized, no limit on daily activities
Clinical Severity | Measured on study Days 3, 5, 8, 11, 15 and 30.
  Measured by National Early Warning Score (NEWS): vital sign based score from 0-20, higher score indicates higher degree of illness
Clinical Severity | Measured on study Days 3, 5, 8, 11, 15 and 30.
  Measured by duration of use of supplemental oxygen (if applicable)
Clinical Severity | Measured on study Days 3, 5, 8, 11, 15 and 30.
  Measured by duration of use of mechanical ventilation (if applicable)
Clinical Severity | Measured on study Days 3, 5, 8, 11, 15 and 30.
  Measured by duration of hospitalization

OTHER OUTCOMES:
Incidence of New Onset Lymphopenia | Through study completion, average of 30 days
  Incidence of new onset lymphopenia during hospitalization measured by blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Conigliaro, MD, Principal Investigator — Northwell Health
Locations (5):
- United States (5):
  - Southside Hospital, Bay Shore, New York
  - North Shore University Hospital, Manhasset, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Lenox Hill Hospital, New York, New York
  - Long Island Jewish Medical Center, Queens, New York

REFERENCES:
- [Background] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Background] Marmor MF, Kellner U, Lai TY, Melles RB, Mieler WF; American Academy of Ophthalmology. Recommendations on Screening for Chloroquine and Hydroxychloroquine Retinopathy (2016 Revision). Ophthalmology. 2016 Jun;123(6):1386-94. doi: 10.1016/j.ophtha.2016.01.058. Epub 2016 Mar 16. PMID 26992838
- [Background] Amrane S, Tissot-Dupont H, Doudier B, Eldin C, Hocquart M, Mailhe M, Dudouet P, Ormieres E, Ailhaud L, Parola P, Lagier JC, Brouqui P, Zandotti C, Ninove L, Luciani L, Boschi C, La Scola B, Raoult D, Million M, Colson P, Gautret P. Rapid viral diagnosis and ambulatory management of suspected COVID-19 cases presenting at the infectious diseases referral hospital in Marseille, France, - January 31st to March 1st, 2020: A respiratory virus snapshot. Travel Med Infect Dis. 2020 Jul-Aug;36:101632. doi: 10.1016/j.tmaid.2020.101632. Epub 2020 Mar 20. PMID 32205269
- [Background] Fox RI. Mechanism of action of hydroxychloroquine as an antirheumatic drug. Semin Arthritis Rheum. 1993 Oct;23(2 Suppl 1):82-91. doi: 10.1016/s0049-0172(10)80012-5. PMID 8278823
- [Background] Yao Y, Tian Y, Zhou J, Ma X, Yang M, Wang S. Epidemiological characteristics of SARS-CoV-2 infections in Shaanxi, China by 8 February 2020. Eur Respir J. 2020 Apr 23;55(4):2000310. doi: 10.1183/13993003.00310-2020. Print 2020 Apr. PMID 32139462
- [Background] Wang L, Gao YH, Lou LL, Zhang GJ. The clinical dynamics of 18 cases of COVID-19 outside of Wuhan, China. Eur Respir J. 2020 Apr 23;55(4):2000398. doi: 10.1183/13993003.00398-2020. Print 2020 Apr. PMID 32139464
- [Background] Geleris J, Sun Y, Platt J, Zucker J, Baldwin M, Hripcsak G, Labella A, Manson DK, Kubin C, Barr RG, Sobieszczyk ME, Schluger NW. Observational Study of Hydroxychloroquine in Hospitalized Patients with Covid-19. N Engl J Med. 2020 Jun 18;382(25):2411-2418. doi: 10.1056/NEJMoa2012410. Epub 2020 May 7. PMID 32379955
- [Background] Magagnoli J, Narendran S, Pereira F, Cummings TH, Hardin JW, Sutton SS, Ambati J. Outcomes of Hydroxychloroquine Usage in United States Veterans Hospitalized with COVID-19. Med. 2020 Dec 18;1(1):114-127.e3. doi: 10.1016/j.medj.2020.06.001. Epub 2020 Jun 5. PMID 32838355
- [Background] Freedberg DE, Conigliaro J, Wang TC, Tracey KJ, Callahan MV, Abrams JA; Famotidine Research Group. Famotidine Use Is Associated With Improved Clinical Outcomes in Hospitalized COVID-19 Patients: A Propensity Score Matched Retrospective Cohort Study. Gastroenterology. 2020 Sep;159(3):1129-1131.e3. doi: 10.1053/j.gastro.2020.05.053. Epub 2020 May 22. No abstract available. PMID 32446698
- [Background] Wang Y, Zhang D, Du G, Du R, Zhao J, Jin Y, Fu S, Gao L, Cheng Z, Lu Q, Hu Y, Luo G, Wang K, Lu Y, Li H, Wang S, Ruan S, Yang C, Mei C, Wang Y, Ding D, Wu F, Tang X, Ye X, Ye Y, Liu B, Yang J, Yin W, Wang A, Fan G, Zhou F, Liu Z, Gu X, Xu J, Shang L, Zhang Y, Cao L, Guo T, Wan Y, Qin H, Jiang Y, Jaki T, Hayden FG, Horby PW, Cao B, Wang C. Remdesivir in adults with severe COVID-19: a randomised, double-blind, placebo-controlled, multicentre trial. Lancet. 2020 May 16;395(10236):1569-1578. doi: 10.1016/S0140-6736(20)31022-9. Epub 2020 Apr 29. PMID 32423584
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343